CLINICAL TRIAL: NCT00432315
Title: Multicenter Phase II Study Evaluating Docetaxel and CDDP as Induction Regimen Prior to Surgery or Radiochemotherapy With Docetaxel, Followed by Adjuvant Docetaxel Therapy in Chemonaive Patients With NSCLC Stage II, IIIa and IIIb
Brief Title: Docetaxel in Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_AT1_203
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Docetaxel

ARMS (2):
- 1 (Experimental): Resectable NSCLC
  Interventions: Drug: Docetaxel + CDDP
- 2 (Experimental): Unresectable NSCSC
  Interventions: Drug: docetaxel + CDDP

INTERVENTIONS:
Drug: Docetaxel + CDDP — * 3 cycles chemotherapy : docetaxel + CDDP
  * Surgery (if no histologically proven R0-resection could be achieved,additional adjuvant radiotherapy should be considered)
  * 3 cycles adjuvant chemotherapy docetaxel
  Arms: 1
Drug: docetaxel + CDDP — * 3 cycles chemotherapy: docetaxel + CDDP
  * Radiochemotherapy
  * 3 cycles adjuvant chemotherapy docetaxel
  Arms: 2

SUMMARY:
Primary objective:

• To assess the response rate to induction therapy with docetaxel/CDDP.

Secondary objectives:

To assess

* Resectability after induction therapy
* Time to progression
* Overall survival
* Safety profile
* Quality of Life

ELIGIBILITY:
Inclusion Criteria:

1. Histology and staging of the disease

   * Histologically or cytologically confirmed NSCLC; histology may include: large cell, squamous cell or adenocarcinoma but no SCLC
   * Resectable or unresectable NSCLC stage II (T1-2 N1, T3 N0) or stage IIIa (T1-2 N2 or T3 N1-2) or stage IIIb (T1-3 N3 or T4 N0-3)
   * Measurable disease (bidimensionally or unidimensionally according to WHO criteria)
2. General conditions

   * Karnofsky Status > 70, if age > 70 years → PS > 70
   * Adequate hematological function (Hb > 10 g/dl, ANC > 2.0 x 109/L, platelets > 100 x 109/L)
   * Adequate renal and hepatic functions: total bilirubin < 1 x upper normal limit (UNL), serum creatinine < 1 x UNL, in case of limit value the creatinine clearance should be > 60 ml/min, ASAT and ALAT < 2.5 x UNL, alkaline phosphatase < 5 x UNL.

Exclusion Criteria:

1. Diagnosis

   * Evidence of brain metastases or other distant metastasis equivalent to stage IV disease
   * History of prior malignancies, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix or other curatively treated cancer with no evidence of disease for at least five years
   * Other serious concomitant illness or medical condition:

     * Congestive heart failure or angina pectoris, except if medically controlled, history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmia
     * History of significant neurologic or psychiatric disorders, including dementia or seizure
     * Active infection requiring i.v. Antibiotics
     * Active ulcer, unstable diabetes mellitus or other contraindications to corticotherapy
   * Hepatic function abnormality: ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL
   * Current peripheral neuropathy WHO grade > 2
2. Prior or concurrent therapy

   * Prior chemotherapy or immunotherapy for NSCLC, including neoadjuvant or adjuvant treatment
   * Prior surgery or radiotherapy for NSCLC
   * Concurrent treatment with other experimental drugs, unapproved medical procedures or other anticancer therapy
3. General conditions

   * Pregnant or lactating patients
   * Patients (M/F) with reproductive potential not implementing adequate contraceptive measurements

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess the response rate to induction therapy with docetaxel in combination with CDDP | every 3 months until tumour progression and thereafter every 6 months until death

SECONDARY OUTCOMES:
Resectability after induction therapy | every 3 months until tumour progression and thereafter every 6 months until death
Time to progression | every 3 months until tumour progression and thereafter every 6 months until death
Overall survival | every 3 months until tumour progression and thereafter every 6 months until death
Safety profile | throughout the study
Quality of life | every 3 months until tumour progression and thereafter every 6 months until death

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Edlmayer, Dr., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Vienna, Austria